CLINICAL TRIAL: NCT00330668
Title: Recombinant Human Insulin-Like Growth Factor-1 (IGF-1) Treatment of Children With Growth Failure Associated With Primary IGF-1 Deficiency: An Open-Label, Multi-Center, Extension Study
Brief Title: Treatment of Children and Adolescents With Growth Failure Associated With Primary IGF-1 Deficiency
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unacceptable frequency of hypoglycemia observed at and above 200 ug/kg/day
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS306; 2019-000844-81 (EudraCT Number)
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Results first posted 2011-06-27 (Estimated); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Growth Disorders
Keywords: Insulin-like Growth Factor Deficiency; IGF-1; Short Stature
MeSH Terms: conditions — Growth Disorders; Dwarfism | interventions — mecasermin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All rhIGF-1 Subjects (Experimental): All subjects entering MS306 began recombinant human insulin-like growth factor-1 (rhIGF-1) twice a day (BID) treatment. Each subject treated in MS301 had an MS306 starting dose that was based on their dose at the completion of MS301 (i.e. subcutaneous injections of rhIGF-1 at 40, 80, or 120 micrograms [μg]/ kilogram [kg] BID).
  MS301 untreated control subjects were randomised in MS306 in a 1:1 ratio to a dose of either 80 or 120 μg/kg rhIGF-1 BID.
  Following Protocol Amendment 1, all subjects received either 80 or 120 μg/kg rhIGF-1 BID until the implementation of Protocol Amendment 2.
  Following Protocol Amendment 2, all subjects were first switched to receive subcutaneous injections of 160 μg/kg rhIGF-1 once a day (QD), followed by individual dose-escalation first to 200 μg/kg rhIGF-1 QD and subsequently to a targeted maximum dose of 240 μg/kg rhIGF-1 QD. Subjects were treated QD until the early termination of the study.
  Interventions: Drug: rh IGF-1 (mecasermin)

INTERVENTIONS:
Drug: rh IGF-1 (mecasermin) — Patients from untreated arm for prior study MS301 (NCT00125164) were randomized to a dose of either 80 or 120 mcg/kg twice daily. For patients receiving active treatment in previous study MS 301 (NCT00125164), they started on a dose of 80 or 120 mcg/kg twice daily based on the dose reached at end of the previous study. Following a protocol amendment in May 2009, all patients were switched to once daily doses of 160 µg/kg, escalated to a targeted maximum dose of 240 µg/kg.
  Other Names: Increlex

SUMMARY:
This is an extension study to Tercica study MS301 (NCT00125164) and is intended to collect long term safety and efficacy data on the continued use of recombinant human insulin-like growth factor-1 (rh IGF-1) in children and adolescents treated for primary IGF-1 deficiency (IGFD). The secondary objective is to use the data collected to learn more about the relationship of IGF-1 exposure to the promotion of normal growth and pubertal development.

DETAILED DESCRIPTION:
Primary IGFD is a term that has been used to describe patients with intrinsic cellular defects in GH action. In this protocol, subjects that have completed one year of mecasermin treatment on Tercica protocol MS301 (NCT00125164) will be allowed to enroll in this extension study. All subjects were planned to receive treatment.

This is a Phase IIIb open-label, multi-center, parallel dose, extension study conducted in approximately 40 centers across the United States.

ELIGIBILITY:
Inclusion Criteria:

* Parents or legally authorized representatives must give signed informed consent before any trial related activities are conducted
* Where required, assent of the subject will be appropriately documented prior to any study related activities
* Completion of assessments at Visit 9 (Month 120 of Study MS301 [NCT00125164])

Exclusion Criteria:

* Incomplete participation in MS301 (NCT00125164)
* Known or suspected allergy to the trial product (mecasermin, recombinant human IGF-1 injection) or its formulation
* Development or presence of a chronic condition except as approved by the Medical Monitor
* Pregnancy
* Any social or medical condition that, in the opinion of the investigator, would be detrimental to either the subject or the study

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2005-11; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr Vice President, Clinical Development and Medical Affairs, Study Director — Ipsen (formerly Tercica, Inc.)
Locations (1):
- Ipsen, Paris, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects that completed study MS301 (NCT00125164) were eligible to enter this Phase 3b, open-label, extension study in prepubertal and pubertal male and female subjects with growth failure associated with primary insulin-like growth factor-1 deficiency (IGFD). This study (MS306) was terminated early by the sponsor on 01 December 2009.
Pre-assignment Details: As subjects entered MS306 whilst MS301 was continuing, dosages were adjusted in MS306 after MS301 data became available. Baseline study data for MS306 were taken from the data collected for Visit 9 (Month 12) of study MS301.
Groups:
- All rhIGF-1 Subjects: All subjects entering MS306 began recombinant human insulin-like growth factor-1 (rhIGF-1) twice a day (BID) treatment. Each subject treated in MS301 had an MS306 starting dose that was based on their dose at the completion of MS301 (i.e. subcutaneous injections of rhIGF-1 at 40, 80, or 120 micrograms [μg]/ kilogram [kg] BID). MS301 untreated control subjects were randomised in MS306 in a 1:1 ratio to a dose of either 80 or 120 μg/kg rhIGF-1 BID.
  Following Protocol Amendment 1, the dosing regimen was changed and all subjects received either 80 or 120 μg/kg rhIGF-1 BID until the implementation of Protocol Amendment 2.
  Following Protocol Amendment 2, all subjects were first switched to receive subcutaneous injections of 160 μg/kg rhIGF-1 once a day (QD), followed by individual dose-escalation first to 200 μg/kg rhIGF-1 QD and subsequently to a targeted maximum dose of 240 μg/kg rhIGF-1 QD. Subjects were treated QD until the early termination of the study.
Period: BID Dosing Period
Arm/Group | All rhIGF-1 Subjects
Started | 114
Completed | 78
Not Completed | 36
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 7
Not completed — Non-Compliance | 5
Not completed — Withdrawal by Subject | 19
Not completed — Sponsor's decision | 1
Not completed — Other | 3
Period: QD Dosing Period
Arm/Group | All rhIGF-1 Subjects
Started | 78
Completed | 0
Not Completed | 78
Not completed — Sponsor decision to terminate study | 74
Not completed — Other | 1
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Groups:
- All rhIGF-1 Subjects: All subjects entering MS306 began rhIGF-1 BID treatment. Each subject treated in MS301 had an MS306 starting dose that was based on their dose at the completion of MS301 (i.e. subcutaneous injections of rhIGF-1 at 40, 80, or 120 μg/kg BID). MS301 untreated control subjects were randomised in MS306 in a 1:1 ratio to a dose of either 80 or 120 μg/kg rhIGF-1 BID.
  Following Protocol Amendment 1, the dosing regimen was changed and all subjects received either 80 or 120 μg/kg rhIGF-1 BID until the implementation of Protocol Amendment 2.
  Following Protocol Amendment 2, all subjects were first switched to receive subcutaneous injections of 160 μg/kg rhIGF-1 QD, followed by individual dose-escalation first to 200 μg/kg rhIGF-1 QD and subsequently to a targeted maximum dose of 240 μg/kg rhIGF-1 QD. Subjects were treated QD until the early termination of the study.
Arm/Group | All rhIGF-1 Subjects
Number analyzed (Participants) | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.5 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 82
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic | 6
  White | 100
  Black | 1
  Asian | 4
  Native Hawaiian | 1
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Height Velocity During BID Dosing Period
Description: Height was measured standing, without shoes, as the average of 3 measurements by the same observer identical technique with a Harpenden or other wall-mounted stadiometer at baseline and each study visit up to 3 years. Height velocity (during any interval of time (annualised) is computed as (height on date 2 - height on date 1)/(age on date 2 - age on date 1) where height is expressed as centimetres so that height velocity is expressed as centimetres per year (cm/yr). Height velocity is presented for subjects completing each year of BID treatment (i.e. Year 1 [0-1 years], Year 2 [1-2 years], Year 3 [2-3 years]).
Time Frame: At Years 1, 2 and 3 in BID dosing period.
Population: The modified Intent-To-Treat (MITT) population included subjects from the ITT population who were randomised to 120 μg/kg rhIGF-1 BID (either in MS301 or MS306). The subjects in the 80 μg/kg group were not analysed for efficacy due to the variations in their dose regimen and the duration of the regimen.
Measure: Mean (Standard Deviation); unit: cm/year
Groups:
- 120 μg/kg rhIGF-1 BID (MITT Population): Subjects in the MITT population received 120 μg/kg rhIGF-1 BID and received the same dose throughout the BID phase of the study.
Arm/Group | 120 μg/kg rhIGF-1 BID (MITT Population)
Number analyzed (Participants) | 55
cm/year
  Year 1: number analyzed (Participants) | 54
  Year 1 | 7.7 (1.5)
  Year 2: number analyzed (Participants) | 44
  Year 2 | 6.1 (1.4)
  Year 3: number analyzed (Participants) | 16
  Year 3 | 5.9 (1.1)

2. Secondary Outcome: Mean Change From Baseline in Height Standard Deviation (SD) Score During BID Dosing Period
Description: Height was measured standing, without shoes, as the average of 3 measurements by the same observer using identical technique with a Harpenden or other wall-mounted stadiometer at baseline and each study visit up to 3 years. Height SD score was determined using the National Center for Health Statistics 2000 data as provided by the Center for Disease Control. The SD score was calculated as the patient value minus the mean divided by the standard deviation. The mean and the standard deviation vary depending on the age and sex of the child. Mean change from baseline in height SD score is presented for all subjects completing each year of BID treatment (i.e. Year 1 [0-1 years], Year 2 [1-2 years], Year 3 [2-3 years]).
Time Frame: At baseline and Years 1, 2 and 3 in BID dosing period.
Population: The MITT population included subjects from the ITT population who were randomised to 120 μg/kg rhIGF-1 BID (either in MS301 or MS306). The subjects in the 80 μg/kg group were not analysed for efficacy due to the variations in their dose regimen and the duration of the regimen.
Measure: Mean (Standard Deviation); unit: SD score/year
Arm/Group | 120 μg/kg rhIGF-1 BID (MITT Population)
Number analyzed (Participants) | 55
SD score/year
  Year 1: number analyzed (Participants) | 54
  Year 1 | 0.5 (0.3)
  Year 2: number analyzed (Participants) | 44
  Year 2 | 0.7 (0.4)
  Year 3: number analyzed (Participants) | 16
  Year 3 | 0.9 (0.6)

3. Secondary Outcome: Mean Change From Baseline in Body Mass Index (BMI) SD Score During BID Dosing Period
Description: BMI SD score was calculated using the National Center for Health Statistics 2000 data as provided by the Center for Disease Control. The SD score was calculated as the patient value minus the mean divided by the standard deviation. The mean and the standard deviation vary depending on the age and sex of the child. Mean change from baseline in BMI SD score is presented for all subjects completing each year of BID treatment (i.e. Year 1 [0-1 years], Year 2 [1-2 years], Year 3 [2-3 years]).
Time Frame: At baseline and Years 1, 2 and 3 in BID dosing period.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SD score/year
Arm/Group | 120 μg/kg rhIGF-1 BID (MITT Population)
Number analyzed (Participants) | 55
SD score/year
  Year 1: number analyzed (Participants) | 54
  Year 1 | 0.3 (0.5)
  Year 2: number analyzed (Participants) | 44
  Year 2 | 0.2 (0.5)
  Year 3: number analyzed (Participants) | 16
  Year 3 | 0.4 (0.5)

4. Secondary Outcome: Mean Change From Baseline in Bone Age During BID Dosing Period
Description: Radiographs of the left hand and wrist were taken on an approximately annual basis for determination of bone (skeletal) age. The films were sent to a central facility for standardised evaluation. Mean change from baseline in bone age is presented for all subjects completing each year of BID treatment (i.e. Year1 [0-1 years], Year 2 [1-2 years], Year 3 [2-3 years]).
Time Frame: At baseline and Years 1, 2 and 3 in BID dosing period.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | 120 μg/kg rhIGF-1 BID (MITT Population)
Number analyzed (Participants) | 55
Years
  Year 1: number analyzed (Participants) | 53
  Year 1 | 1.2 (0.5)
  Year 2: number analyzed (Participants) | 38
  Year 2 | 2.3 (0.6)
  Year 3: number analyzed (Participants) | 12
  Year 3 | 3.4 (0.7)

5. Secondary Outcome: Mean Change From Baseline in Predicted Adult Height During BID Dosing Period
Description: Predicted adult heights were estimated using the Roche-Wainer-Theissen method which takes into account changes in age, height and bone age. Mean change from baseline in predicted adult height is presented for all subjects completing each year of BID treatment (i.e. Year 1 [0-1 years], Year 2 [1-2 years], Year 3 [2-3 years]).
Time Frame: At baseline and Years 1, 2 and 3 in BID dosing period.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | 120 μg/kg rhIGF-1 BID (MITT Population)
Number analyzed (Participants) | 55
cm
  Year 1: number analyzed (Participants) | 53
  Year 1 | 2.7 (2.0)
  Year 2: number analyzed (Participants) | 38
  Year 2 | 3.9 (3.2)
  Year 3: number analyzed (Participants) | 12
  Year 3 | 3.7 (3.4)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the overall study (including both the BID and QD dosing periods) from Day 1 until early termination of the study (up to 4 years, 3 months).
Description: The safety population included all subjects who received at least one dose of study medication.
Groups:
- All rhIGF-1 Subjects: All subjects entering MS306 began recombinant human insulin-like growth factor-1 (rhIGF-1) BID treatment. Each subject treated in MS301 had an MS306 starting dose that was based on their dose at the completion of MS301 (i.e. subcutaneous injections of rhIGF-1 at 40, 80, or 120 μg/kg BID).
  MS301 untreated control subjects were randomised in MS306 in a 1:1 ratio to a dose of either 80 or 120 μg/kg rhIGF-1 BID.
  Following Protocol Amendment 1, all subjects received either 80 or 120 μg/kg rhIGF-1 BID until the implementation of Protocol Amendment 2.
  Following Protocol Amendment 2, all subjects were first switched to receive subcutaneous injections of 160 μg/kg rhIGF-1 QD, followed by individual dose-escalation first to 200 μg/kg rhIGF-1 QD and subsequently to a targeted maximum dose of 240 μg/kg rhIGF-1 QD. Subjects were treated QD until the early termination of the study.
Arm/Group | All rhIGF-1 Subjects
All-Cause Mortality (participants affected / at risk) | 0/114
Serious Adverse Events (participants affected / at risk) | 6/114
Other Adverse Events (participants affected / at risk) | 107/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All rhIGF-1 Subjects (N=114)
Appendicitis (Infections and infestations) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Forearm Fracture (Injury, poisoning and procedural complications) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Otitis Externa (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All rhIGF-1 Subjects (N=114)
Abdominal Pain Upper (Gastrointestinal disorders) | 20 (27)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (15)
Arthropod Bite (Injury, poisoning and procedural complications) | 7 (7)
Blood Glucose Decreased (Investigations) | 7 (8)
Bronchitis (Infections and infestations) | 8 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (27)
Diarrhoea (Gastrointestinal disorders) | 13 (13)
Dizziness (Nervous system disorders) | 6 (7)
Ear Infection (Infections and infestations) | 10 (13)
Ear Pain (Ear and labyrinth disorders) | 7 (9)
Gastroenteritis (Infections and infestations) | 9 (14)
Gastroenteritis Viral (Infections and infestations) | 20 (23)
Headache (Nervous system disorders) | 35 (86)
Hypoglycaemia (Metabolism and nutrition disorders) | 46 (72)
Influenza (Infections and infestations) | 22 (31)
Influenza Like Illness (General disorders) | 9 (18)
Injection Site Bruising (General disorders) | 9 (10)
Injection Site Hypertrophy (General disorders) | 16 (30)
Lymphadenopathy (Blood and lymphatic system disorders) | 8 (8)
Molluscum Contagiosum (Infections and infestations) | 7 (7)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 7 (13)
Nasopharyngitis (Infections and infestations) | 22 (34)
Otitis Externa (Infections and infestations) | 11 (16)
Otitis Media (Infections and infestations) | 20 (28)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 10 (13)
Pharyngitis Streptococcal (Infections and infestations) | 23 (32)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 14 (21)
Pyrexia (General disorders) | 28 (43)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Seasonal Allergy (Immune system disorders) | 6 (6)
Sinusitis (Infections and infestations) | 12 (24)
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 8 (11)
Upper Respiratory Tract Infection (Infections and infestations) | 38 (79)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 8 (10)
Vomiting (Gastrointestinal disorders) | 23 (44)

LIMITATIONS AND CAVEATS:
The study was terminated by the sponsor due to an unacceptably high incidence of hypoglycaemia observed in approximately 50% of the subjects receiving 200 μg/kg rhIGF-1 or greater QD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each investigator may publish or report data from their own subjects. The trial data in aggregate are the property of Tercica, Inc. and may not be published without permission of Tercica, Inc. Tercica, Inc. will be the final arbitrator of issues relating to the publication or presentation of the aggregate data.